CLINICAL TRIAL: NCT02894229
Title: The Mindfulness Intervention and Repeated Acute Stress (MIRAS) Study
Brief Title: The Stress Reduction Intervention Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Ohio University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16F18
Record Dates: First submitted 2016-09-05; First posted 2016-09-09 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Stress, Physiological; Stress, Psychological
MeSH Terms: conditions — Stress, Psychological | interventions — Mindfulness-Based Stress Reduction; Cognitive Behavioral Therapy; Population Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- No intervention wait-list (No Intervention): This arm will receive no intervention for approximately the first 4 months. At the conclusion of the 4-month period, this group will receive a 6-week cognitive-behavioral therapy (CBT) group
- Mindfulness Based Stress Reduction(MBSR) (Active Comparator): This arm will receive 6 weekly, 2-hour groups that focuses on mindfulness meditation for stress reduction
  Interventions: Behavioral: Mindfulness Based Stress Reduction
- Cognitive Behavioral Therapy (CBT) Group (Active Comparator): This are will receive 6 weekly, 2-hour groups that focus on cognitive-behavioral skills for stress
  Interventions: Behavioral: Cognitive-Behavioral Therapy (CBT) Group

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction — A modified version of traditional MBSR. The current study's version of MBSR is shortened to 6-weeks.
  Arms: Mindfulness Based Stress Reduction(MBSR)
Behavioral: Cognitive-Behavioral Therapy (CBT) Group — A 6-week, 2-hour per group, skills group that focuses on various cognitive-behavioral skills for stress reduction (e.g., progressive muscle relaxation; cognitive restructuring).
  Arms: Cognitive Behavioral Therapy (CBT) Group

SUMMARY:
The primary purpose of the present study is to investigate the relationship between mindfulness and stress habituation. The investigators propose to measure the effect of mindfulness on stress habituation by randomly assigning participants to a 6-week mindfulness-based stress reduction group intervention, a cognitive-behavioral skills group comparison intervention, or a waitlist control condition followed by repeated acute psychosocial stress testing (2 laboratory sessions on 2 separate days). Saliva will be collected from participants throughout both laboratory testing sessions to measure HPA axis activation (an essential stress-responsive system), along with other measures of physiological and psychological stress (e.g., heart rate, blood pressure, emotions). Mediators and moderators of treatment outcome will be examined. The cognitive-behavioral skills group condition is an appropriate comparison group due to the well-documented efficacy of cognitive-behavioral interventions on stress.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking adults who are between the ages of 18-50, who are in general good health
* Perceived stress scores (PSS) > 3 on a screening survey

Exclusion Criteria:

* reported previous completion of a Mindfulness-Based Stress Reduction or Cognitive Behavioral Therapy program.
* reported pregnancy
* reported use of steroid medication
* presence of a major psychiatric or endocrine disorder (e.g., Major Depression, Cushings Disease; self-reported)
* reported regular wake time after 10:00 AM on a weekday

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale | Baseline and 6-weeks after baseline.
  A 10-item self-report measure that examines perceived stress. The measure produces one total score. The investigators will measure the change in total score from baseline to the 6-week assessment.
Salivary cortisol response to repeated acute psychosocial stress | Post-intervention (approximately 7-14 weeks after baseline assessment)
  4 saliva samples will be collected before and after a psychosocial stressor task, which will be administered on two separate occasions separated in time by at least 48 hours. All saliva samples will be assayed for salivary cortisol using enzyme-linked immunoassays. The investigators will measure the change in cortisol stress profiles from the first stressor exposure to the second.

SECONDARY OUTCOMES:
Cardiovascular response to repeated acute psychosocial stress | Post-intervention (approximately 7-14 weeks after baseline assessment)
  Heart rate and blood pressure will be assessed non-invasively and periodically before, during, and after non-invasively a psychosocial stressor task, with an Omron Health Care HEM-907XL Professional Blood Pressure Monitor. The investigators will measure the change in heart rate and blood pressure stress profiles from the first stressor exposure to the second.
Autonomic response to repeated acute psychosocial stress | Post-intervention (approximately 7-14 weeks after baseline assessment)
  Heart rate variability will be assessed continuously before, during, and after non-invasively a psychosocial stressor task, with a MP150 device manufactured by BIOPAC. The investigators will measure the change in heart rate variability stress profiles from the first stressor exposure to the second.
Dispositional Mindfulness | Baseline and 6-weeks
  Five Facet Mindfulness Questionnaire
Equanimity | Baseline and 6-weeks
  The Non-Attachment Scale
Smoking | Baseline and 6-weeks
  Fagerstrom Test for Nicotine Dependence
Alcohol | Baseline and 6-weeks
  Alcohol Use Disorders Identification Test - Consumption items
Marijuana | Baseline and 6-weeks
  Single item assessing frequency of marijuana use
Perceived control over thoughts | Baseline and 6 weeks
  Thought Control Ability Questionnaire
Coping Skills | Baseline and 6-weeks
  Brief-COPE measure
Depressed mood | Baseline and 6-weeks
  Center for Epidemiologic Studies Depression Scale
Anxiety | Baseline and 6-weeks later
  Spielberger State-Trait Anxiety Inventory
Social Connectedness | Baseline and 6-weeks
  Social Connectedness Scale-Revised
Optimism | Baseline and 6-weeks
  Life Orientation Test
Worry | Baseline and 6-weeks
  Penn State Worry Questionnaire
Experiential Avoidance | Baseline and 6-weeks
  Acceptance and Action Questionnaire-II
Emotion Regulation | Baseline and 6-weeks
  Difficulties in Emotion Regulation Scale
Negative Urgency | Baseline and 6-weeks
  UPPS-P Impulsive Behavior Scale: Negative Urgency Items
Chronic Stress | Baseline and 6-weeks
  Trier Inventory for Chronic Stress
Sleep | Baseline and 6-weeks
  Pittsburgh Sleep Quality Index
State Affect | Post-intervention (approximately 7-14 weeks after baseline assessment)
  Positive and Negative Affect Schedule (PANAS) will be used to assess state affect and specific emotions several times before and after a psychosocial stressor task. The investigators will measure the change in emotion response profiles from the first stressor exposure to the second.
State mindfulness | Post-intervention (approximately 7-14 weeks after baseline assessment)
  Mindful Attention Awareness Scale (MAAS) - state version. The investigators will measure the change in state mindfulness from the first stressor exposure to the second.
Implicit association between self and shame | Post-intervention (approximately 7-14 weeks after baseline assessment)
  A shame experience and self implicit association test will be used to measure experiential self-referential processing of present moment shame. The investigators will measure the change in implicit association between self and shame from the first stressor exposure to the second.
State rumination | Post-intervention (approximately 7-14 weeks after baseline assessment)
  Thoughts Questionnaire (TQ). The investigators will measure the change in state rumination from the first stressor exposure to the second.
Stress appraisals | Post-intervention (approximately 7-14 weeks after baseline assessment)
  Cognitive task appraisals will be assessed before and after a psychosocial stressor task. The investigators will measure the change in appraisals from the first stressor exposure to the second.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Manigault AW, Shorey RC, Decastro G, Appelmann HM, Hamilton KR, Scanlin MC, France CR, Zoccola PM. Standardized stress reduction interventions and blood pressure habituation: Secondary results from a randomized controlled trial. Health Psychol. 2021 Mar;40(3):196-206. doi: 10.1037/hea0000954. PMID 33630641